CLINICAL TRIAL: NCT01824407
Title: A Double-Blind, Multi-center, Randomized, Sham-Controlled, Parallel Group Comparison of the dermaPACE® (Pulsed Acoustic Cellular Expression) Device in Conjunction With Standard of Care Versus Standard of Care Alone in the Treatment of Diabetic Foot Ulcers
Brief Title: A Comparison of the dermaPACE® (Pulsed Acoustic Cellular Expression) Device in Conjunction With Standard of Care Versus Standard of Care Alone in the Treatment of Diabetic Foot Ulcers
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: SANUWAVE, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SAN12-DERM02
Record Dates: First submitted 2013-04-01; First posted 2013-04-04 (Estimated); Last update posted 2014-03-06 (Estimated); Status verified 2014-03

CONDITIONS: Diabetic Foot Ulcers
Keywords: foot; ulcers; diabetes; wound; healing
MeSH Terms: conditions — Diabetic Foot; Ulcer; Diabetes Mellitus; Wounds and Injuries

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Active device plus standard of care (Active Comparator): Active device plus standard of care
  Interventions: Device: Electrohydraulic-generated shock wave
- Sham device plus standard of care (Sham Comparator): dermaPACE device that uses a dummy applicator that does not emit shock waves
  Interventions: Device: Sham device plus standard of care

INTERVENTIONS:
Device: Electrohydraulic-generated shock wave
  Other Names: dermaPACE
  Arms: Active device plus standard of care
Device: Sham device plus standard of care
  Arms: Sham device plus standard of care

SUMMARY:
The Sponsor of this study, SANUWAVE, Inc., has developed an investigational device known as the dermaPACE® (Pulsed Acoustic Cellular Expression) device for the possible treatment of diabetic foot ulcers. This device generates acoustic (sound) pressure waves designed to act on the cells in your body to generate proteins that may lead to wound closure. The dermaPACE® device has not been approved for the treatment of diabetic foot ulcers; therefore its use in this study is investigational.

The purpose of the study is to evaluate the ability of the dermaPACE® device to help diabetic foot ulcers heal more quickly. The active study device, the dermaPACE®, will be compared to an inactive look-alike device (called a "Sham") in this study. The sham device will not provide any treatment to your diabetic foot ulcer.

ELIGIBILITY:
Inclusion Criteria:

1. Is >=22 years of age at Visit 1;
2. If female of child-bearing potential, both of the following must be met at Visit 1:

   * Practices one of the following methods of contraception and continues through the duration of the study: hormonal contraceptives, IUD, spermicide and barrier or implantable device, and
   * Has a negative urine qualitative beta-HCG pregnancy test;
3. If female and post-menopausal one of the following must be met at Visit 1:

   * Has had a complete hysterectomy, bilateral salpingo-oophorectomy or tubal ligation or otherwise be incapable of pregnancy, or
   * Is postmenopausal for at least one year;
4. Has at least one DFU that is located in the ankle area or below that has persisted a minimum of 30 days prior to Visit 1.
5. Has Type I or Type II Diabetes Mellitus with a HbA1c <= 11% at Visit 1;
6. Is capable of wound care at home;
7. Has a target ulcer >= 1.0 cm2 and <= 16 cm2 at Visits 1 and 2;
8. Has a target ulcer that is Grade 1 or 2, Stage A according to the University of Texas Diabetic Wound Classification system, at Visits 1 and 2
9. In the leg with the target ulcer has an ABI >= 0.70 and <= 1.20 OR if the ABI is >1.20 has a toe pressure >50 mmHg OR tcpO2 > 40 mmHg at Visit 1;
10. Subject agrees, or if applicable, the subject's legal representative agrees that the subject can participate in the study

Exclusion Criteria:

1. Is currently pregnant or plans to become pregnant during the study;
2. Is nursing or actively lactating;
3. Is morbidly obese (Body Mass Index >= 40) at Visit 1;
4. Has clinically significant renal disease defined as having an estimated creatinine clearance of <=40mL/min at Visit 1;
5. Has osteomyelitis in the foot or ankle on which the target ulcer is located at Visit 1 or 2;
6. Has evidence of a prior ulcer in the same area as the target ulcer;
7. Has a target ulcer that has decreased in volume by 50% or more at Visit 2 as compared to the volume at Visit 1;
8. Has multiple foot ulcers that are connected by fistulas or has an ulcer(s) that are within 5 cm of the target ulcer at Visit 1 or 2;
9. Has a target ulcer that tunnels into wound tracks which cannot be fully visualized from the wound surface at Visit 1 or 2;
10. Has active cellulitis either at the site of, or in the surrounding area of, the target ulcer at Visit 1 or 2;
11. Has a target ulcer that has visually purulent exudates or that has malodorous exudates on examination at Visit 1 or 2;
12. Has PVD, per Doppler Ultrasound, requiring vascular surgery intervention at Visit 1 or 2;
13. Requires use of off-loading Diabetic Walker device for the foot intended for study application for a reason other than for a target ulcer on the plantar surface of the foot at Visit 1 or 2;
14. Has had a lower extremity revascularization procedure within eight weeks of Visit 1;
15. Has active Charcot foot at Visit 1 or 2;
16. Has had a surgical procedure to correct biomechanical abnormities within eight weeks of Visit 1;
17. Has had a deep vein thrombosis within six months of Visit 1;
18. Has clinical evidence of lymphedema at Visit 1;
19. Has had chemotherapy within 60 days of Visit 1;
20. Has a life expectancy <=2 years;
21. Has previously participated in a dermaPACE diabetic foot ulcer study;
22. Has had treatment of the target ulcer with growth factors, prostaglandin therapy, negative pressure or vasodilator therapy within two weeks of Visit 1;
23. Is receiving >=10 mg/day of steroid therapy;
24. Has sickle cell anemia;
25. Has a known immunodeficiency disorder to include, but not be limited to: AIDS, HIV, etc.
26. Has received radiation treatment within 120 days of Visit 1;
27. Has received treatment with immunosuppressants within sixty days of Visit 1;
28. Has received treatment with biologically active cellular products on the target ulcer, e.g. Apligraf®, Dermagraft®, etc. within sixty days of Visit 1;
29. Has received treatment with acellular (collagen-based) products on the target ulcer, e.g. Alloderm®, Integra®, etc. within 30 days of Visit 1;
30. Has a current history of substance abuse (current is defined as within 120 days of Visit 1);
31. Has a history of major systemic infections requiring hospitalization within three months of Visit 1 ;
32. Has a current malignancy or a history of malignancy within five years, of Visit 1 except for basal cell carcinoma that has been treated with local excision and is no longer present;
33. Has a physical or mental disability or geographical concerns that would inhibit compliance with required study visits;
34. Is planning to undergo an exclusionary treatment or procedure during the study; or
35. Has participated in another investigation within 30 days of Visit 1

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2013-03; Primary Completion 2014-04 (Estimated)

PRIMARY OUTCOMES:
Complete closure | 12 weeks
  Complete closure will be assessed by visual inspection by the principal or sub-investigator according to the following complete closure definition: 100% skin re-epithelializion without drainage or dressing requirements confirmed at two consecutive study visits. A re-epithelialized target ulcer is defined as the tissue surface having at least a thin layer of epithelium covering the prior, previously denuded, target ulcer area.

SECONDARY OUTCOMES:
Volumetric reduction | 12 weeks
  Digital planimetry will be used to assess volumetric reduction between follow-up visits.
Area reduction | 12 weeks
  Digital planimetry will be used to assess area reduction between follow-up visits.
Rate of recurrence | 24 weeks
Rate of amputation and other adverse events | 24 weeks

CONTACTS AND LOCATIONS:
Locations (19):
- United States (18):
  - Associated Foot and Ankle Specialists, Phoenix, Arizona
  - Southern Arizona VA Healthcare System, Tucson, Arizona
  - Long Beach VA Healthcare System, Long Beach, California
  - Foot and Ankle Clinic, Los Angeles, California
  - Alameda County Medical Center - Highlands Campus, Oakland, California
  - Lucius J. Hill DPM, San Bernardino, California
  - Paul and Margaret Brand Research Center at Barry University, Hialeah, Florida
  - The Research Center, Hialeah, Florida
  - River City Clinical Research, Jacksonville, Florida
  - St. Paul Medical Research, Miami, Florida
  - Advanced Pharma CR, Miami, Florida
  - Northwestern University, Div of Plastic and Reconstructive Surgery, Chicago, Illinois
  - Foot Healthcare Associates, Southfield, Michigan
  - Moore Foot and Ankle Specialists, Asheville, North Carolina
  - Wound Center - ACMH, Kittaning, Pennsylvania
  - Podiatric Medical Partners of Texas, Dallas, Texas
  - UT Southwestern Medical Center, Dallas, Texas
  - Foot and Ankle Associates of SW Virginia, Roanoke, Virginia
- The Mayer Institute, Hamilton, Ontario, Canada